CLINICAL TRIAL: NCT00234845
Title: A Multi-Centre Randomized, Double-Blind Study Comparing Adalimumab (D2E7) Plus Methotrexate With Placebo Plus Methotrexate on Work Disability in Subjects With Early Rheumatoid Arthritis
Brief Title: Adalimumab in Combination With Methotrexate vs Methotrexate Alone in Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-527
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adalimumab
Drug: methotrexate

SUMMARY:
The purpose of the study is to evaluate the effectiveness of adalimumab in combination with methotrexate compared to methotrexate alone on work disability in subjects with early rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 or older and in good health (Investigator discretion) with a recent stable medical history
* Subject has a diagnosis of rheumatoid arthritis as defined by the 1987-revised ACR criteria
* Subject must be in paid employment
* Subject has self-reported work impairment since onset of symptoms

Exclusion Criteria:

* A subject has chronic arthritis diagnosed before age 16 years.
* Subject has been on preceding treatment with methotrexate Subject unable to withdraw from current DMARDs
* Subject has preceding treatment with any biological TNF antagonist
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-03

PRIMARY OUTCOMES:
Job loss measurement

SECONDARY OUTCOMES:
Job productivity measurements
Patient reported outcomes
DAS28
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, Abbott Park, Illinois, United States

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778